CLINICAL TRIAL: NCT05840354
Title: Repetitive Transcranial Magnetic Stimulation Combined with Steroid Joint Injection for the Treatment of Chronic Spinal Pain: Protocol for a Pilot Randomized Controlled Trial
Brief Title: RTMS and Steroid Joint Steroid Injection in Chronic Spinal Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Western University, Canada (Other); St. Joseph's Health Care London (Other)
Responsible Party: Principal Investigator, Siobhan Schabrun, Professor and William and Lynne Gray Research Chair in Mobility and Activity, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SJIrTMS
Record Dates: First submitted 2023-04-04; First posted 2023-05-03 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Chronic Spinal Pain
Keywords: repetitive transcranial magnetic stimulation; steroid joint injection; inflammatory markers; inflammation; chronic pain
MeSH Terms: conditions — Inflammation; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active repetitive transcranial magnetic stimulation + steroid joint injection (Active Comparator): Active transcranial stimulation will be delivered for a total of 11 sessions. Each session will consist of 40 trains of 5s delivered at 10 Hz, at an intensity of 85% of the resting motor threshold for the first dorsal interosseous muscle and an intertrain interval of 25s (total of 2000 stimulations in a 20-minute session).
  Interventions: Device: Magstim Rapid2
- sham repetitive transcranial magnetic stimulation + steroid joint injection (Sham Comparator): The sham repetitive transcranial magnetic stimulation coil will be delivered using a Placebo D70mm Air Film Coil of identical colour, size, and shape as the active rTMS coil. The sham coil uses a magnetic shield that blocks the magnetic field from being delivered to the scalp while producing a similar auditory click during discharge. All other aspects of the rTMS protocol will be identical between the active and sham conditions.
  Interventions: Device: Placebo D70mm Air Film Coil

INTERVENTIONS:
Device: Magstim Rapid2 — 1-4 weeks after administration of the SJI, participants will attend their first rTMS session. rTMS will be delivered using a biphasic stimulator (DuoMag) and a figure-of-eight coil to the corticomotor representation of the first dorsal interosseous muscle contralateral to the side of worst pain. Recording electrodes will be positioned in a belly-tendon montage over the FDI for electromyography recording. The hotspot and resting motor threshold (rMT) of the FDI will be determined and saved using a Brainsight Neuronavigation system to ensure accurate coil repositioning within and between sessions.
  The hotspot and rMT will be confirmed and adjusted if needed at each intervention session. Each rTMS session will consist of 40 trains of 5s delivered at 10Hz, at an intensity of 85% of the resting motor threshold for the FDI muscle and an intertrain interval of 25s (total of 2000 stimulations in a 20-minute session).
  Other Names: rTMS
  Arms: active repetitive transcranial magnetic stimulation + steroid joint injection
Device: Placebo D70mm Air Film Coil — Sham intervention will follow same protocol as active rTMS using a sham coil that does not deliver actual magnetic stimulation.
  Other Names: sham rTMS
  Arms: sham repetitive transcranial magnetic stimulation + steroid joint injection

SUMMARY:
Chronic spinal pain (CSP) is one of the most common chronic pain conditions globally. Steroid joint injections (SJI) are a routine treatment option for patients with CLBP that is recalcitrant to other treatments. However, SJI has been shown to have limited long-term efficacy with patients often requiring another injection within months to adequately control pain. One option to prolong the analgesic effects of SJI is to use a type of noninvasive brain stimulation called repetitive transcranial magnetic stimulation (rTMS). Previous studies have shown rTMS may be capable of providing long-term pain relief in patients with chronic back pain. However, the literature on rTMS in patients with CSP is limited and no study has explored rTMS in patients receiving recurrent SJI for pain control.

In this pilot randomized controlled trial study, we'll be investigating if combining rTMS with SJI in CSP individuals will enhance or prolong the analgesic effects of SJI alone.

The investigators hypothesize that a combined rTMS and SJI intervention will be feasible, tolerable, and safe and will have larger and longer-lasting effects on CSP than a sham rTMS and SJI intervention.

DETAILED DESCRIPTION:
Background:

Chronic spinal pain (CSP) is one of the most common health conditions globally. The pathophysiology of CSP is complex, and it is thought that a spectrum of peripheral and central mechanisms may be involved. (Baron et al., 2016) Steroid joint injections (SJI) are a routine therapeutic intervention for patients with CSP that is recalcitrant to other types of treatment. However, SJI has been shown to have limited long-term efficacy with patients requiring another injection within months to adequately control pain (Won et al., 2020). One option to prolong the analgesic effects of SJI may be to incorporate repetitive transcranial magnetic stimulation (rTMS) as an adjunct therapy. Studies have shown rTMS may be capable of providing long-term pain relief in patients with CSP (Ambriz-Tututi et al., 2016). However, the literature on rTMS in patients with CSP is limited and no study has explored rTMS in patients receiving concurrent SJI for pain control.

Thus, the aims of this study are to determine: (1) the feasibility, tolerability, safety, and perceived patient response to a combined rTMS and SJI intervention, and (2) whether rTMS combined with SJIs (active rTMS group) display trends towards greater benefits for pain and function than SJIs alone (sham rTMS group). We hypothesize that a combined rTMS and SJI intervention be feasible, tolerable, and safe and will show trends towards larger and longer-lasting effects on chronic spinal pain than a sham rTMS and SJI intervention.

Study Design:

This pilot study is a randomized, participant- and assessor-blind controlled trial of active and sham repetitive transcranial magnetic stimulations (rTMS) in a population of individuals with CSP, who are receiving recurrent SJIs at three- to six-month intervals through the St Joseph's Pain Clinic. The rTMS intervention will begin 1-4 weeks after SJI and include a 2-week induction phase with active or sham rTMS delivered 3 times each week. The purpose of the induction phase is to strengthen the effects of rTMS at the start of the treatment through multiple sessions in a relatively short period of time. A maintenance phase will follow and in weeks 3, 4, 6, 8, and 12 participants will receive a single active or sham rTMS session. Pain severity will be assessed weekly using an electronic diary from baseline (the week of SJI until week 24). Disability and quality of life will be assessed at baseline, 4, 8, 12, 18 and 24 weeks.

Participants:

Forty adults (≥18 years old) with CSP who are currently receiving recurrent SJIs for control of CLBP at the St. Joseph's Health Centre Pain Clinic in London, Ontario, Canada will be recruited.

Sample Size:

This is a pilot randomized controlled study designed to generate data that can be used to inform a future large-scale trial should the intervention appear feasible, safe and show trends of effectiveness. Thus, the investigators have selected a sample size of 20 individuals per group for a total of 40 participants. A sample size of 40 participants was selected as this is considered achievable within the time frame allocated for the completion of the pilot study according to participant recruitment rates within the pain clinic. The aim is to evaluate key trial parameters, such as recruitment and retention of participants, randomization, the success of blinding, acceptability of the intervention, levels of missing data and preliminary indications of effectiveness, to inform the calculation of a sample size for powering a full trial.

Steroid Joint Injections (SJI):

SJI will be given by an interventional pain physician following the standard clinical procedure for the St. Joseph's Health Centre Pain Clinic. The treatment team will determine how many joints will be injected based on their standard clinical assessment.

Repetitive transcranial magnetic stimulation (rTMS):

1-4 weeks after SJI administration, participants will attend their first rTMS session. Electromyography (EMG) electrodes will be placed in a belly-tendon montage over the first dorsal interosseous (FDI) muscle, with the specific side (left or right) chosen based on the participant's side with the worst CSP. A Brainsight Neuronavigation system will coordinate a Magstim Rapid2 stimulator and its D70mm Remote Control Stimulating Coil accessory on the cranium to identify and save the hotspot and resting motor threshold (rMT) of the FDI, targeting the corticomotor representation contralateral to the side of worst CSP. This setup ensures precise coil positioning. The hotspot and rMT will be confirmed and adjusted if needed at each intervention session to maintain accuracy and safety.

Following this setup, rTMS will be delivered to the FDI muscle representation using the same Magstim Rapid2 stimulator but with a different coil, the D70mm Air Film Coil, on the side contralateral to the worst CSP. Each rTMS session will consist of 40 trains of 5s delivered at 10Hz, at an intensity of 85% of the resting motor threshold for the FDI muscle and an intertrain interval of 25s (total of 2000 stimulations in a 20-minute session). Previous studies have used a similar protocol in chronic back pain and shown that a minimum of 1000 stimulations of high-frequency rTMS is necessary to produce a significant reduction in the outcome measures for pain, and disability (Cruccu et al., 2016).

Sham rTMS will be delivered using a Placebo D70mm Air Film Coil of identical colour, size, and shape as the active rTMS coil. The sham coil uses a magnetic shield that blocks the magnetic field from being delivered to the scalp while producing a similar auditory click during discharge. All other aspects of the rTMS protocol will be identical between the active and sham conditions.

Confidentiality and Data Security:

All study data will be stored electronically on the institutional REDCap database, and within the hospital network. Access to study data and/or medical records will be limited to authorized study personnel only. A master log with identifiers will be stored as a password-protected document on the hospital's secure network, separately from the study data.

The participant will be able to withdraw at any point during data collection. The data will be unable to be withdrawn once it has been pooled with other participants' data for statistical tests for the purposes of a paper or abstract however these data will be de-identified.

Statistical Analysis:

All statistical analyses will be carried out using the software R. Data for feasibility and safety will be analyzed using descriptive statistics. To determine trends of effectiveness, analyses of pain and disability will be performed according to intention-to-treat and per protocol using analysis of variance (ANOVA) to assess change within groups and the differences between groups over time (pre/post). All data will be assessed for normality using the Shapiro-Wilk test. Normally distributed data will be assessed using 2-way repeated measures of ANOVA with 2 levels for intervention (active rTMS/sham rTMS) and levels for time (0, 4, 8, 12, and 24 weeks) as separate factors. If significant group x time interactions are found, then Bonferroni post hoc tests will be used to determine which means are significantly different from one another. Non-parametric data will be assessed via a Mann-Whitney U test on change scores between groups. The effect size will be determined using partial η2 from planned contrasts. The size of the treatment effects will be used to determine whether it is worthwhile to conduct a full randomized controlled trial in the future. Given the pilot nature of this trial, missing data will not be replaced. Bonferroni post hoc tests will be applied if appropriate. The α will be set at 0.05 for all tests.

Results will be corrected for false discovery rate using Benjamini-Hochberg correction where an adjusted p-value of < 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Currently receiving recurrent steroid joint injections for control of chronic spinal pain at the St. Joseph's Health Centre Pain Clinic in London, Ontario, Canada,
* Have pain in the spinal region of an intensity ≥4 out of 10 in the week before your most recent steroid joint injection,
* Have received at least 2 steroid joint injections within the last 12 months at regular intervals
* Have had a consistent medication regimen for the past 3 months.

Exclusion Criteria:

* Unable to read, understand, and speak English and are not able to give consent
* Known or suspected serious spinal pathology (tumour, fracture, dislocation, scoliosis)
* Spinal surgery in the past 12 months
* History of uncontrolled mental health condition(s)
* Meet any specific rTMS-related exclusion criteria listed on the safety screening questionnaire (S1; Rossi et al., 2008).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Measures of feasibility and tolerability | Through study completion, an average of 24 weeks
  Data for feasibility, tolerability, and safety will be analyzed using descriptive statistics. Feasibility and tolerability will be measured as (1) the time taken to complete the recruitment of 40 participants, (2) the number of sessions attended by each participant, (3) the number of dropouts in each group, (4) the proportion of participants recruited from the total number screened, and (5) the willingness of each participant to undergo therapy on an 11-point numerical rating scale with 'not at all willing' at 0 and 'very willing' at 10 (measured at baseline).
Measures for safety | Through study completion, an average of 24 weeks
  Safety will be presented as any adverse reaction reported on verbal questioning at each session. The assessor will record a description of any adverse reactions along with the severity, duration and how the adverse reaction was managed. The number of participants reporting adverse reactions, and the duration and severity of the adverse reactions will be reported.

SECONDARY OUTCOMES:
Pain Numeric Rating Scale | Weeks 1 through 24
  Pain severity will be assessed at baseline and weekly until week 24 using the 11-point Pain Numeric Rating Scale.
Brief Pain Inventory - Short Form (BPI-SF) | Weeks 4, 8, 12, 24
  Pain severity and the impact of pain on the patient's daily functioning will be assessed using the 9-item, Brief Pain Inventory short form at baseline, weeks 4, 8, 12, and 24.
12-Item Short Form (SF-12) | Weeks 4, 8, 12, 24
  The 12-item short form (SF-12) will be used to assess the quality of life and will be taken at baseline, weeks 4, 12 and 24.
Oswestry Disability Index (ODI) | Weeks 4, 8, 12, 24
  Disability will be assessed using the Oswestry Disability Index (ODI) at baseline, weeks 4, 8, 12, and 24. The 12-item short form (SF-12) will be used to assess the quality of life and will be taken at baseline, weeks 4, 12 and 24. Finally, as rTMS has previously been shown to positively affect depression and anxiety symptoms, the Depression Anxiety and Stress Scale 21 (DASS-21) will be used to monitor any potential effects our rTMS treatment has on mood. This will be administered at weeks 4, 12, and 24.
Global Rating of Change Scale (GRC) | Weeks 4 - 24
  A 15-point GRC, with -7 "a very great deal worse", 0 "about the same", to 7 "a very great deal better", will be administered to assess participants' perception of symptom improvement or worsening in response to treatment. The GRC will be administered in weeks 4, 12 and 24.
Depression Anxiety and Stress Scale 21 (DASS-21) | Weeks 4, 12, 24
  As rTMS has previously been shown to positively affect depression and anxiety symptoms, the Depression Anxiety and Stress Scale 21 (DASS-21) will be used to monitor any potential effects our rTMS treatment has on mood. This will be administered at weeks 4, 12, and 24.

CONTACTS AND LOCATIONS:
Overall Officials: Siobhan Schabrun, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (2):
- Canada (2):
  - St. Joseph's Health Care London, London, Ontario
  - Parkwood Institute (Main Building), London, Ontario

IPD SHARING:
Plan to Share IPD: No